CLINICAL TRIAL: NCT06681740
Title: CARDIOINSPIRE - Effectiveness of Adding Inspiratory Muscle Training to a Cardiac Rehabilitation Program for People With Ischemic Heart Disease Revascularized by Percutaneous Transluminal Coronary Angioplasty.
Brief Title: Effectiveness of Inspiratory Muscle Training for People With Ischemic Heart Disease Revascularized by Percutaneous Transluminal Coronary Angioplasty.
Acronym: CARDIOINSPIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Jose Maria Zuazagoitia de la Lama-noriega, University professor. Graduate in Physiotherapy. Master in New Trends in Health Sciences Research., University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SICEIA-2024-001869
Record Dates: First submitted 2024-10-31; First posted 2024-11-08 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Myocardial Ischemia; Coronary Arterial Disease (CAD)
Keywords: Myocardial Ischemia; Coronary Arterial Disease (CAD); Inspiratory Muscle Training; Cardiac Rehabilitation
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training group (Experimental): The intervention group will be given an inspiratory muscle training device that will be regulated at 70% of their Maximum Inspiratory Pressure. This load is able to induce improvements in their musculature.
  Interventions: Device: Inspiratory muscle training
- Control group (Sham Comparator): The control group will be given an inspiratory muscle training device that will be regulated with a load of 5 cm H2O. This load is not sufficient to induce changes in the musculature, so it will function as a placebo.
  Interventions: Device: Sham Inspiratory muscle training

INTERVENTIONS:
Device: Inspiratory muscle training — The control group will perform a standard cardiac rehabilitation program, consisting of 16 multicomponent exercise sessions, health education, and a weekly group of psychological therapy session. The intervention group will do the same program with the addition of Inspiratory Muscle Training (IMT). The following device will be used: Power Breath model: Medic Classic. The training will be performed by adjusting the device load to 70% of the Maximum Inspiratory Pressure value, performing 1 daily training session 4 days a week of 3 sets of 10 repetitions, with a rest of 3 minutes between sets, during 8 weeks. A physical therapist will teach participants how to use the device on the first day and they will be instructed to perform it at home. They will be given a diary to record their compliance. In addition, once a week the physiotherapist will supervise the execution of the IMT by the participants.
  Other Names: IMT
  Arms: Inspiratory muscle training group
Device: Sham Inspiratory muscle training — The control group will be given the same device as experimental group, but the load for all of the participants of the control group will be 5cm de H2O. This load is so low that it´s not able to induce improvement of the inspiratory musculature.
  Other Names: Sham
  Arms: Control group

SUMMARY:
Myocardial Ischemia (MI) consists of the narrowing of the internal lumen of the arteries that perfuse the heart. As the section of the artery decreases, so does the blood flow and therefore the supply of oxygen to the myocardium, which can cause angina pectoris or even an acute myocardial infarction. It is the leading cause of death from cardiovascular disease, responsible for 9.44 million deaths in 2021 and 185 million disability-adjusted life years. For this reason, it is one of the most important public health problems in all countries in the world that entails high health and social spending.

The non-pharmacological strategy with the most evidence currently to improve the quality of life of patients and also prevent subsequent cardiovascular events are cardiac rehabilitation programs (CRP). These include smoking cessation, control of other cardiovascular risk factors, health education, psychological therapy and a multimodal exercise program. Two types of exercise are performed, cardiovascular or aerobic resistance and strength. There is limited evidence on the addition of inspiratory muscle training (IMT) in people with MI. For this reason, it is not routinely recommended in clinical practice guidelines. Therefore, this thesis project, based on a clinical trial, tries to increase knowledge on this topic.

In view of the above, the main objective of this project is to analyze the effectiveness of adding inspiratory muscle training to a CRP of people with ischemic heart disease revascularized by percutaneous transluminal coronary angioplasty (PTCA) after 16 intervention sessions, based on to functional capacity, in addition to muscle strength, social support, anxiety, depression, coping with the disease, sexual dysfunction, quality of life, quality of sleep, eating habits and body composition. On the other hand, the secondary objectives are to know the biopsychosocial profile of this population and analyze gender differences through a subgroup analysis.

To achieve these objectives, a low-risk randomized and controlled clinical trial will be carried out in parallel at the Virgen de la Victoria University Hospital in Málaga (HUVV). People from this health area diagnosed with MI who have undergone PTCA will be recruited. The control group will complete the usual 8-week cardiac rehabilitation program with 2 weekly sessions of multicomponent exercise (cardiovascular and strength), one weekly session of health education and another of group psychological therapy. The intervention group will do the same program to which an IMT will be added. It will be performed with loads of 70% of the Maximum Inspiratory Pressure (MIP) value, completing 3 sets of 10 repetitions, 4 days a week, with 3 minutes of rest between sets, during the 8 weeks that the PRC lasts. Different measurements will be made and various tests and questionnaires will be passed before and after the PRC and the effect of adding or not adding the IMT on the variables to be analyzed will be analyzed using statistical methods.

It is expected that some of the variables will improve since there is some evidence (low and moderate) of this, as concluded by a recent review. Furthermore, in similar clinical populations such as patients with heart failure (HF), there is a high level of evidence that several of these parameters improve. Therefore, it can be expected that the results are similar in MI. In those variables without prior evidence, we hypothesize that there will be an improvement, since increasing MIP in isolation has been shown, in different clinical populations, to improve the functional capacity and quality of life of the study subjects.

If the expected benefits are finally observed, the current evidence on the use of IMT in CRPs for people with MI and PTCA will increase. In anticipation of the accumulated evidence of the effectiveness of the proposed treatment, the results derived from the present study may recommend including the IMT as another fundamental component of the CRP for this subgroup of patients.

DETAILED DESCRIPTION:
Myocardial ischemia According to the Spanish Heart Foundation, myocardial ischemia (MI) is the disease caused by atherosclerosis of the coronary arteries, responsible for providing blood to the heart muscle. Coronary atherosclerosis is a slow process of collagen formation and accumulation of lipids (fats) and inflammatory cells (lymphocytes) that causes narrowing of the lumen of the coronary arteries. This process begins in the first decades of life, but does not present symptoms until the stenosis of the coronary artery becomes so severe that it causes an imbalance between the supply of oxygen to the myocardium and its metabolic needs3. In this case, myocardial ischemia occurs, which may be chronic, known as chronic coronary syndrome or stable angina pectoris, or sudden occlusion due to thrombosis of the artery, which causes a lack of oxygenation of the myocardium that gives rise to coronary syndrome. Acute also called unstable angina and acute myocardial infarction. MI reduces force production, causes arrhythmias, and causes muscle damage, leading to acute ischemic contractile failure of the heart. Patients with chronic ischemic heart disease have lower evaluations of their social life and their coping with daily routine.

The consequence of the processes described above is that people who suffer from MI decrease their tolerance to exercise, functionality and performance in activities of daily living, which leads them to sedentary behaviors, worsening their quality of life. Furthermore, a vicious circle of inactivity and clinical and functional deterioration is established that produces a general worsening of physical condition and atrophy of peripheral and respiratory muscles. All of these circumstances lead to a decrease in functional capacity and therefore to a worse prognosis of the disease.

Regarding the risk factors that lead to the development of MI, there is a combination of socioeconomic, metabolic, behavioral and environmental risk factors. Among them are advanced age, high blood pressure, an unhealthy diet, high cholesterol, diabetes, obesity, smoking, a sedentary lifestyle, stress, family history and harmful consumption of toxins, among others. Most of these factors are modifiable and it is one of the fundamental pillars of their treatment to get affected people to change their lifestyle. The incidence is higher in men since women benefit from a hormonal protective effect during their fertile life. This circumstance disappears with menopause, which equalizes the cases in both sexes from 45-50 years of age.

Epidemiology It is estimated that in 2020 there were 244.1 million people living with MI worldwide. Of them, 141 million were men and 103.1 million were women. The regions of North Africa, the Middle East, Central Asia, South Asia and Eastern Europe had the highest prevalence rates. The global mortality rate was 112.37 per 100,000, this being also higher in the regions with the highest prevalence.

MI affects approximately 126 million people worldwide, representing 1.72% of the world's population. It is the main cause of death, with 9 million deaths annually. The incidence begins to increase in the fourth decade of life and is higher in men than in women. In developed countries, about a third of all deaths in people over 35 years of age are attributed to this disease. In the United States, it is estimated that almost half of men and approximately one-third of women will experience some symptoms of MI during their lifetime. In the European Union, cardiovascular diseases account for 40% of all deaths. Furthermore, the economic costs associated with MI are significant. The treatment of cardiovascular diseases constitutes 54% of total health expenditure, and contributes approximately a quarter of productivity losses.

Coronary heart disease is closely related to aging. Therefore, despite the decrease in its incidence observed in recent decades, all indicators suggest that its incidence will increase in the years to come. Coronary syndromes are expected to increase between 69% and 119% by 2049, mainly due to the growth of the population of patients over 75 years of age. For the group of patients between 25 and 75 years of age, the incidence is projected to remain stable in the coming decades.

Treatment

It usually consists of thrombolysis (revascularization of the artery or arteries whose flow is compromised) and can be done in two ways:

* By open surgery performing a bridge between two vessels that redirects blood to the affected myocardium.
* By performing a percutaneous transluminal coronary angioplasty (PTCA). This option is less invasive and uses a balloon at the tip of a thin tube, called a catheter, to widen the artery. A small spring is usually placed to keep the artery open.

Secondary prevention Once the first cardiovascular event has occurred, it is important to prevent it from happening again. This is called secondary prevention. In this regard, the non-pharmacological strategy with the most evidence at present to reduce mortality, cardiovascular disability, improve the quality of life of patients and prevent further cardiovascular events is cardiac rehabilitation programs (CRP). Moreover, their cost-effectiveness is well known. These include smoking cessation, control of other cardiovascular risk factors, health education, psychological therapy, and a multimodal exercise program (cardiovascular and strength training). Usually 2-3 training sessions are performed weekly for 8-10 weeks.

Inspiratory muscle training Specific inspiratory muscle training (IMT) consists of applying higher than usual workloads to the muscles responsible for generating the necessary negative pressure inside the thorax for air to enter the lungs. This overload induces adaptations that produce an increase in the strength of this musculature. It is widely used as part of the treatment of people with chronic respiratory diseases and people with heart failure (HF). It is a very safe intervention that reduces dyspnea and improves functional capacity and quality of life in these patients.

Overload is achieved by breathing in through specific devices containing a valve whose threshold can be regulated. In order to decide the pressure at which each individual will train, his or her Maximum Inspiratory Pressure (MIP) must be measured beforehand. Training protocols at high loads, between 50% and 80% of the MIP, are those that obtain the best results according to the available evidence for patients with HF and for patients revascularized with grafting by open surgery. Therefore, the intervention will be performed with loads of 70% of the MIP value, completing 3 sets of 10 repetitions, 4 days a week, with 3 minutes rest between sets, during the 8 weeks of the CRP.

Hypothesis and Objectives

Justification In view of the perspective presented above and the available literature, it is pertinent to conduct a low-risk randomized clinical trial evaluating the effectiveness of the addition of IMT to a CRP of people with IC with PTCA. A recently published review9 concludes that the quality of the evidence for inspiratory muscle training for the improvement of maximal oxygen consumption and expiratory muscle strength in this population is very low. However, it should be taken into account that most of the clinical trials carried out to date have been performed on patients who underwent open surgery, so that the literature is scarce in percutaneously operated patients. In this sense, the results of our study will be specifically focused on percutaneously revascularized patients, thereby increasing knowledge of the effects of this intervention in the subgroup of patients with IHD and PTCA on these and other variables. Although CRP have been shown to be effective there is limited evidence on the addition of an IMT in patients with IHD. Clinical practice guidelines do not routinely recommend IMT due to this lack of evidence, so we aim to shed light on its effectiveness.

Hypotheses The addition of inspiratory muscle training to a cardiac rehabilitation program for people with percutaneously revascularized ischemic heart disease will lead to better results in terms of functional capacity and muscle strength, in addition to social support, anxiety, depression, coping with the disease, sexual dysfunction, quality of life, quality of sleep, eating habits and body composition, after 16 sessions of intervention compared to the control group.

H2.- It is expected that a large proportion of the participants will present anxiety and depression, poor coping with the disease and poor control of cardiovascular risk factors.

H3.- There will be greater effects of the intervention on the variables in the subgroup of women, due to their greater degree of commitment to the intervention program.

Objectives

I. General objective

- To analyze the effectiveness of the addition of inspiratory muscle training to a cardiac rehabilitation program in people with percutaneously revascularized ischemic heart disease after 16 sessions of intervention, based on functional capacity, in addition to muscle strength, social support, anxiety, depression, coping with the disease, sexual dysfunction, quality of life, sleep quality, eating habits and body composition.

II. Secondary objectives

* To know the biopsychosocial profile of this population based on functional capacity, in addition to muscular strength, social support, anxiety, depression, coping with the disease, sexual dysfunction, quality of life, quality of sleep, eating habits and body composition.
* To analyze gender differences through subgroup analysis. Methodology

The present clinical trial has been previously approved by the Provincial Research Ethics Committee of Malaga with Code SICEIA-2024-001869 in its session number 9, held on 09/26/2024.

The characteristics of the proposed clinical trial are reported in accordance with the SPIRIT standards (Standard Protocol Items: Recommendations for Interventional Trials).

Study design Randomized, controlled (parallel), triple-blind, low-risk clinical trial.

Study Setting The study will be carried out at the Cardiac Rehabilitation Unit (CRU) of the Hospital Universitario Virgen de la Victoria de Málaga (HUVV).

Study Subjects Persons with Myocardial Ischemia (MI) referred to the CRU of the HUVV who have undergone PTCA.

Inclusion criteria: i) people with MI with PTCA; ii) both sexes; iii) over 18 years of age; iv) under 80 years of age; v) absence of cognitive deficit and/or physical limitations that would prevent them from performing physical exercise or completing the questionnaires necessary for participation in the study.

Exclusion criteria: i) Disease or condition that contraindicates exercise such as severe hypertrophic obstructive cardiomyopathy, severe aortic stenosis and/or dissecting aortic aneurysm; ii) Patients who refuse treatment or do not sign the informed consent.

Sampling, Sample Size and Randomization Consecutive sampling will be carried out with patients attending the HUVV CRU and meeting the criteria described above.

The sample size was calculated to detect differences between groups in our main variable, functional capacity measured by maximal oxygen consumption. According to the meta-analysis by Fabero-Garrido et al , people with ischemic heart disease who have undergone an inspiratory muscle training program have a mean difference of 2.18 ml O2/kg/min with respect to the control group and we want to find a deviation of 1 MET (3.5 ml O2/kg/min). The calculations were carried out with the statistical software G*Power 3.1, considering in all cases a confidence level of 95% and a power of 80%.

In view of the above, a sample size of 33 subjects per group (66 in total) was established. In addition, to minimize the impact of possible dropouts, the total sample was increased by 10% to 72 patients, which will lead to the final inclusion of 36 patients in each group.

Randomization of participants will be performed through a computer program that generates a sequence of random numbers.

Cardiac Rehabilitation Program.

The usual CRP will be carried out and supervised by the usual multidisciplinary team of the HUVV. It is composed of a cardiologist, a rehabilitation physician, a physiotherapist, a nurse and a psychologist. Prior to inclusion in the study, each participant will undergo a simple ergometry test to determine their maximum heart rate (MHR), observe their behavior at maximum effort and rule out conditions that contraindicate exercise. The study subjects will attend the cardiac rehabilitation room of the hospital 3 days a week. Two of these days will be dedicated to physical exercise sessions and the third to health education and a group psychological therapy session.

The health education session will deal with a different topic each week (basic knowledge of their pathology, proper medication, safe physical exercise, sexual dysfunction, healthy eating and control of cardiovascular risk factors).

On the other hand, those subjects suffering from erectile dysfunction will be offered the possibility of being seen in the urology office. The rehabilitation physician will perform a nutritional assessment by bioimpedanciometry and a morphological assessment of the quadriceps and another of abdominal fat, both by ultrasound. Participants with poorly controlled diabetes and/or morbid obesity will see the endocrinologist of the cardiac rehabilitation team.

The training sessions will last approximately 75 minutes. The structure will be as follows:

* Reception of patients, taking of constants (blood pressure, heart rate and glycemia in case of diabetic patients) and placement of telemetry.
* Warm up
* Strength Exercise: It will consist of different exercises with dumbbells and elastic bands involving various joints. We will work at 50% of 1 repetition maximum (1RM) measured indirectly with the method of 20 repetitions maximum (20RM). Three sets of 10 repetitions of the following exercises will be completed: elbow flexion, shoulder abduction and knee extension. The rest interval between sets will be 30 seconds.
* Cardiovascular Exercise: It will be performed on a treadmill or stationary bicycle. It will have a duration of 30 minutes. The first month the patient will be trained at 70% of the heart rate resulting from applying the Karvonen formula and the second month at 80%. The modality may be continuous or intervallic depending on the patient's tolerance.
* Relaxation and return to calm: patients will remain seated in chairs for 5 minutes during which a guided relaxation audio will be played.
* Checking of constants and farewell.

Patients will be weighed every week to monitor their evolution and rule out possible adverse effects of the training. The program will be extended for 8 weeks until completing 16 concurrent training sessions. At the end of the program, ergometry, blood analysis and the rest of the tests will be repeated.

Masking

None of the participants will know to which group they belong since they will all be given the same EEMI device. For the control group a load of 5 cmH2O will be set. This work intensity is below that necessary to achieve adaptations in the inspiratory muscles and will therefore function as a placebo.

The evaluators will also not know to which group the study subjects belong since they will not participate in the assignment or intervention process.

The analysis will be done independently since the data will be delivered coded.

Statistical analysis

Measures of central tendency and dispersion will be used for numerical variables, as well as relative frequencies for categorical variables to assess comparability between groups. All relevant variables will be examined for this purpose.

Exploratory data analysis will be performed to identify and address outliers that may affect the results. Appropriate corrections will be applied to mitigate their influence.

To contrast the differences between the control and experimental groups, the Student's t-test for independent samples or the nonparametric Mann-Whitney test will be used according to the normality of the data, measured with the Kolmogorov-Smirnov test. For pre- and post-intervention comparisons, Student's t test for paired samples will be used in case of normality or the Wilcoxon test, otherwise. In the case of qualitative variables, chi-square test will be used.

In addition to the aforementioned statistical analyses, possible complex and nonlinear relationships between variables will be explored by means of regression models or multivariate analyses, such as multiple regression or principal component analysis.

The analyses will be performed with the IBM SPSS v.24 statistical program. Anticipated risks and contingency plans

Anticipated risk Contingency plan:

Non-compliance of participants with the IMT Submission of paper log of compliance in the form of a diary

Incorrect performance of the IMT technique Weekly reinforcement session at HUVV

Doubts about the performance of the IMT by the participants The physiotherapist supervising the CRP physical exercise will always be available during the sessions to clarify any doubts.

Prospective It would be interesting to study in future clinical trials the specific training of the expiratory musculature (EMT) in these patients, both in isolation and concurrently with inspiratory training. There are studies that have shown benefits in postural stability and walking speed due to the strengthening of the central musculature of the body.

It would also be interesting to measure the medium- and long-term effects of EMT, as so far existing studies have not done so.

Justification of available resources The University of Cadiz, through its Library, will provide the bibliographic resources necessary for the development of this research project, such as access to the main publishers and indexed scientific journals.

The HUVV will provide the facilities and materials used by the CRP for this study.

The interviews and some of the pre- and post-intervention measurements will be carried out in the cardiac rehabilitation office of the HUVV. Its dimensions are 7m2 and it has the following materials:

* JAMARTm approved hydraulic dynamometer.
* Hogan Health Industries hand-held dynamometer, MicroFet 2 model.
* Measuring tape.
* Bioimpedance meter, Akern brand, Nutrilab model.
* MicroRPM® digital portable manometer.

Physical training, health education sessions, group psychology therapies and some measurements will be carried out in the cardiac rehabilitation room of the HUVV. It has an area of 80m2. and has the following equipment:

* 2 treadmills.
* 6 exercise bikes.
* Dumbbells.
* Elastic bands.
* Telemetry systems for patients.
* Computer with the necessary software to monitor electrocardiograms and heart rates (Mortaraâ system).
* Monitors where to observe the electrography in real time.
* Chairs for taking constants and for health education and relaxation sessions.
* Loudspeaker and playback system for relaxation audios.
* Blood pressure monitors, stethoscopes and glucometers to monitor patients' vital signs.
* Defibrillator and stretcher in case of adverse effects.
* 43" flat screen for health education sessions.

Ergometry tests will be performed by a cardiologist and a specialized nurse from the cardiology service of the HUVV in its exercise physiology laboratory. The laboratory is equipped with the following elements:

* Treadmill
* Sphygmomanometer, glucometer and phonendoscope.
* Computer with the appropriate software to perform the incremental exercise protocol.
* Defibrillator.
* Stretcher

This project is supported theoretically and technically by the TIC-256 Intelligent Social Knowledge Based Systems (IntellSOK) research group and the Pain Observatory of the University of Cadiz. Both entities have extensive experience in the development of research studies and have the technical resources and knowledge necessary for the proper implementation of the proposed project.

Ethical and/or biosafety implications of the proposed research. The present project will follow the ethical principles established for medical research on human subjects according to the Declaration of Helsinki.

The present clinical trial has been previously approved by El Comité de Ética e Investigación con medicamentos (CEIm) Provincial de Málaga (Spain), with communication/application code: SICEIA-2024-001869.

Since data from real subjects will be used, it is essential to guarantee their confidentiality, privacy and data protection. To this end, the participation of the subjects will be voluntary, and it is an indispensable requirement to sign the informed consent form for participation in the study. Participants will be able to withdraw from the study whenever they wish to do so. To safeguard the identity of the subjects, their names and surnames will be coded in the database.

This is a low-intervention clinical trial, since IMT is a very safe intervention, as it is routinely performed in other populations of chronic cardiac and respiratory patients without any relevant adverse effects having been reported.

In addition, patients will be scrupulously stratified according to their cardiovascular risk and the cardiac rehabilitation team at the HUVV has extensive experience in training this type of patient and its professionals are in constant training.

The damages incurred by the participants will be covered by the individual or collective self-insurance that the researcher in question has already contracted for the usual practice of his or her profession.

To publish the results of the project in international peer-reviewed journals and present the results at congresses worldwide, the Consolidated Standards of Reporting Trials (CONSORT) statement will be followed. In addition, as part of the knowledge translation strategy, we will disseminate the results on institutional websites and social media, contact news organizations and identify partner institutions interested in the results.

ELIGIBILITY:
Inclusion Criteria:

* people with Myocardial Ischemia and percutaneous transluminal coronary angioplasty
* both sexes
* over 18 years old
* under 80 years of age
* absence of cognitive deficits and/or physical limitations that would prevent them from performing physical exercise or completing the questionnaires required for participation in the study.

Exclusion Criteria:

* disease or condition that contraindicates exercise such as severe hypertrophic obstructive cardiomyopathy
* severe aortic stenosis and/or dissecting aortic aneurysm
* patients who refuse treatment or do not sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Functional Capacity | First measurement between recruitment and the beginning of the intervention, second measurement between the end of the intervention and 2 weeks after the intervention.
  To assess functional capacity, a simple exercise stress test will be performed following the recommendations of the Spanish Society of Cardiology in which the maximum oxygen consumption (VO2max). Ergometry, also known as stress test, is not only a diagnostic technique that analyzes the response of the heart to exercise, but also a test that is able to quantify the oxygen consumption of the individual who performs it. In this study it will be performed on a treadmill. The Bruce protocol will be used, which progressively increases the speed of the treadmill and its inclination every 3 minutes. It will be performed by a cardiologist of the unit. VO2max will be obtained in METS (a metabolic equivalent 1 MET = 3.5 ml O2/kg/min).

SECONDARY OUTCOMES:
The Charlson Comorbidity Index | Between recruitment and the start of intervention
  The Charlson Comorbidity Index, a tool validated in Spanish that evaluates life expectancy at 10 years, will be calculated. It includes 19 items that, if present, have been shown to specifically affect the subject's life expectancy. It was initially adapted to assess one-year survival, but was finally adjusted to assess 10-year survival.
Sleep Quality | First measurement between recruitment and the beginning of the intervention, second measurement between the end of the intervention and 2 weeks after the intervention.
  To assess sleep quality, the Pittsburgh Sleep Quality Index (PSQI) will be used. It is the most widely used self-report questionnaire for this purpose. It consists of 19 self-assessed questions whose overall rating ranges from 0 to 21. Higher scores represent poorer sleep quality. Above 5 is considered a "bad sleeper" and below 5 a "good sleeper". A change of 3 points is the minimum clinically significant difference.
Level of physical activity | First measurement between recruitment and the beginning of the intervention, second measurement between the end of the intervention and 2 weeks after the intervention.
  The level of physical activity will be assessed using the RAPA (RapidAssessmentof Physical Activity) questionnaire validated in Spanish. It was designed to measure this variable in older adults. It consists of 9 items, seven of which seek to determine whether people comply with the recommendation to perform 30 minutes or more of moderate physical activity at least 5 days a week. The two additional items measure whether people perform flexibility and strength exercises. Based on the total score, it establishes the following categories of physical activity: "Sedentary", "Not very active", "Not very active regular light", "Not very active regular" and "Active".
The left ventricular ejection fraction (LVEF) | First measurement between recruitment and the beginning of the intervention, second measurement between the end of the intervention and 2 weeks after the intervention.
  The left ventricular ejection fraction (LVEF) will be measured by the cardiologist by ultrasound following the recommendations of the American Society of Echocardiography for use in clinical trials and also in agreement with expert cardiologists.
Maximal Inspiratory Pressure (MIP) | First measurement between recruitment and the beginning of the intervention, second measurement between the end of the intervention and 2 weeks after the intervention.MIP will be reassessed midway through the program to readjust the training load.
  To measure MIP , the MicroRPM® digital portable manometer (Vyaire Medical GmbH, Hoechberg, Germany) will be used. The assessments of MIP will be performed according to the recommendations of the American Thoracic Society (ATS) and the European Respiratory Society (ERS) and following the protocol of the Spanish Society of Pneumology and Thoracic Surgery (SEPAR). Inspiratory muscle weakness will be considered with values below 62 cmH2O for women and 83 cmH2O for men. MIP will be reassessed midway through the program (at the end of week 4) to readjust the training load.
Maximal Expiratory Pressure (MEP) | First measurement between recruitment and the beginning of the intervention, second measurement between the end of the intervention and 2 weeks after the intervention.
  To measure Maximal Expiratory Pressure (MEP), the MicroRPM® digital portable manometer (Vyaire Medical GmbH, Hoechberg, Germany) will be used. The assessments of PEM will be performed according to the recommendations of the American Thoracic Society (ATS) and the European Respiratory Society (ERS) and following the protocol of the Spanish Society of Pneumology and Thoracic Surgery (SEPAR). Expiratory muscle weakness will be considered with values below 81 cmH2O in women and 109 cmH2O in men.
Quality of life | First measurement between recruitment and the beginning of the intervention, second measurement between the end of the intervention and 2 weeks after the intervention.
  To assess quality of life, the SF-12 questionnaire version 2 (SF-12v2), translated into Spanish and validated in the population of Catalonia, will be administered. It consists of 12 questions, around 8 dimensions: general self-perception of health, physical capacity, physical functioning, emotional role, social functioning, mental health, physical pain and self-perception of vitality with options. It measures 2 main components, physical health (PCS) and mental health (MSC). PCS and MCS scores are standardized on a scale from 0 to 100, where 50 is the mean for the general population. Higher scores indicate better quality of life.
Anxiety and Depression | First measurement between recruitment and the beginning of the intervention, second measurement between the end of the intervention and 2 weeks after the intervention.
  Anxiety and depression will be assessed using the Hospital Anxiety and Depression Scale (HADS), composed of 14 questions, is divided into two subdimensions: anxiety (HADS-A) and depression (HADS-D). Each question has Likert-type responses, with scores ranging from 0 to 3. Thus, each subscale has a score ranging from 0 to 21 points. Scores between 0 and 7 indicate the absence of depression and/or anxiety, scores between 8 and 10 suggest a clinically significant disorder, and scores between 11 and 21 indicate the presence of moderate to severe depression and/or anxiety.
Functional Social Support | First measurement between recruitment and the beginning of the intervention, second measurement between the end of the intervention and 2 weeks after the intervention.
  The Duke scale in its Spanish version will be used to assess functional social support. It is a self-administered questionnaire, with a Likert-type response scale (1-5). The range of scores goes from 11 to 55 points. The score obtained reflects perceived support rather than actual support. The lower score means less support. A score of 32 or more indicates widespread social support, whereas a score of less than 32 indicates low perceived social support.
Erectile Dysfunction | First measurement between recruitment and the beginning of the intervention, second measurement between the end of the intervention and 2 weeks after the intervention.
  To assess erectile dysfunction in male participants, the International Index of Erectile Function in its reduced version (IIEF-5) and validated in Spanish will be used. It is a 5-question self-assessment questionnaire that addresses aspects such as confidence in achieving erections, rigidity of erections, ability to maintain an erection during sexual intercourse, and satisfaction with sexual intercourse. Each question is answered on a scale of 1 to 5, where 5 is the highest score and 1 is the lowest. The total score is obtained by adding the scores of each question, with a range of 5 to 25. It allows to classify erectile dysfunction as mild (17-21), moderate (12-16) or severe (5-11).
Dyspnea | First measurement between recruitment and the beginning of the intervention, second measurement between the end of the intervention and 2 weeks after the intervention.
  To establish the severity of dyspnea, the scale created by the New York Heart Association (NYHA) will be used. It reflects the patient's capacity for physical exertion and is therefore also called "NYHA functional class", which has 4 grades indicating greater dyspnea to a greater degree.
Body Composition by Bioimpedance | First measurement between recruitment and the beginning of the intervention, second measurement between the end of the intervention and 2 weeks after the intervention.
  Bioimpedance will be used to determine the body composition of the participants. It works by sending a mild electrical current through the body and measuring the resistance exerted by the various tissues as it passes through, which varies according to their water and fat content. The measurement will be made with the Akern bioimpedance meter, Nutrilab model. In addition, the body mass index (BMI) of each individual will be calculated after weighing and measuring them in the training room.
Waist circumference | First measurement between recruitment and the beginning of the intervention, second measurement between the end of the intervention and 2 weeks after the intervention.
  The waist circumference will also be measured at the navel with a tape measure.
Nutritional Ultrasound | First measurement between recruitment and the beginning of the intervention, second measurement between the end of the intervention and 2 weeks after the intervention.
  A nutritional ultrasound will be performed. The FujiFilm Sonosite SII ultrasound scanner will be used. The subcutaneous fat in the quadriceps without contraction, the thickness of the rectus femoris muscle (anteroposterior distance), its transverse diameter, its area in cm2 and its circumference will be measured. The thickness of the vastus intermedius will be measured (anteroposterior distance).
  In the abdomen without contraction, total subcutaneous fat, superficial subcutaneous fat and pre-peritoneal fat will be measured.
Eating habits | First measurement between recruitment and the beginning of the intervention, second measurement between the end of the intervention and 2 weeks after the intervention.
  Eating habits will be evaluated by means of the Mediterranean diet adherence questionnaire. It consists of 14 direct questions on the consumption of the main foods of the Mediterranean diet, such as: olive oil, fruits, vegetables, legumes, fish, nuts, wine and white meats. The scores are grouped into four categories: high adherence (12-14 points), medium adherence (8-11.99 points), low adherence (0-7.99 points).
Maximum static quadriceps muscle strength | First measurement between recruitment and the beginning of the intervention, second measurement between the end of the intervention and 2 weeks after the intervention.
  Maximum static quadriceps muscle strength will be measured with the patient seated on a stretcher and the knee flexed at 90º using the Hogan Health Industries model MicroFet 2 hand-held dynamometer.
Hand grip strength | First measurement between recruitment and the beginning of the intervention, second measurement between the end of the intervention and 2 weeks after the intervention.
  Hand grip strength will be measured with a JamarTm approved hydraulic dynamometer. Isometric strength of the hand and forearm muscles will be assessed with the arm extended along the body by performing a contraction for at least 3 seconds. Three maneuvers will be performed at least 20 seconds apart. The highest value obtained will be considered.
Incidents | During the intervention
  During the entire procedure, all incidents that occur, whether cardiological events or not, will be monitored and recorded. They will be analyzed and if they are attributable to the intervention, the corresponding measures will be taken.
The number of sessions | During intervention
  The number of sessions attended by each participant will be taken into account as another variable for the statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Antonio Moral Muñoz, MSc, Phd, Study Director — University of Cadiz; Jose Maria Zuazagoitia de la Lama-Noriega, MSc, PhD student, Principal Investigator — University of Cadiz; Adela Maria Gomez Gonzalez, PhD, Medical Doctor, Study Director — Hospital Universitario Virgen de la Victoria
Locations (1):
- Hospital Universitario Virgen de la Victoria, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No
This is sensitive data that will be processed only in the development of this study.

REFERENCES:
- [Background] Bjarnason-Wehrens B, Predel HG. Inspiratory muscle training - an inspiration for more effective cardiac rehabilitation in heart failure patients? Eur J Prev Cardiol. 2018 Nov;25(16):1687-1690. doi: 10.1177/2047487318798917. Epub 2018 Sep 10. No abstract available. PMID 30198748
- [Background] Lee K, Park D, Lee G. Progressive Respiratory Muscle Training for Improving Trunk Stability in Chronic Stroke Survivors: A Pilot Randomized Controlled Trial. J Stroke Cerebrovasc Dis. 2019 May;28(5):1200-1211. doi: 10.1016/j.jstrokecerebrovasdis.2019.01.008. Epub 2019 Jan 31. PMID 30712955
- [Background] Yamamoto S, Matsunaga A, Wang G, Hoshi K, Kamiya K, Noda C, Kimura M, Yamaoka-Tojo M, Masuda T. Effect of balance training on walking speed and cardiac events in elderly patients with ischemic heart disease. Int Heart J. 2014;55(5):397-403. doi: 10.1536/ihj.14-017. Epub 2014 Aug 4. PMID 25088580
- [Background] Martinez-Gonzalez MA, Garcia-Arellano A, Toledo E, Salas-Salvado J, Buil-Cosiales P, Corella D, Covas MI, Schroder H, Aros F, Gomez-Gracia E, Fiol M, Ruiz-Gutierrez V, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Munoz MA, Warnberg J, Ros E, Estruch R; PREDIMED Study Investigators. A 14-item Mediterranean diet assessment tool and obesity indexes among high-risk subjects: the PREDIMED trial. PLoS One. 2012;7(8):e43134. doi: 10.1371/journal.pone.0043134. Epub 2012 Aug 14. PMID 22905215
- [Background] Garcia-Almeida JM, Garcia-Garcia C, Vegas-Aguilar IM, Ballesteros Pomar MD, Cornejo-Pareja IM, Fernandez Medina B, de Luis Roman DA, Bellido Guerrero D, Breton Lesmes I, Tinahones Madueno FJ. Nutritional ultrasound(R): Conceptualisation, technical considerations and standardisation. Endocrinol Diabetes Nutr (Engl Ed). 2023 Mar;70 Suppl 1:74-84. doi: 10.1016/j.endien.2022.11.010. PMID 36935167
- [Background] Hernández Tatiana Thieme R, Araos F, Hernández RS. Adaptación y Análisis Psicométrico de la Versión Española del Índice Internacional de Función Eréctil (IIEF) en Población Adaptation and Psychometric Analysis of the Spanish Version of the International Index of Erectile Function in Chilean Population. 2017;35:223-30.
- [Background] de la Revilla Ahumada L, Bailon E, de Dios Luna J, Delgado A, Prados MA, Fleitas L. [Validation of a functional social support scale for use in the family doctor's office]. Aten Primaria. 1991 Oct;8(9):688-92. Spanish. PMID 16989055
- [Background] Broadhead WE, Gehlbach SH, de Gruy FV, Kaplan BH. The Duke-UNC Functional Social Support Questionnaire. Measurement of social support in family medicine patients. Med Care. 1988 Jul;26(7):709-23. doi: 10.1097/00005650-198807000-00006. PMID 3393031
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Schmidt S, Vilagut G, Garin O, Cunillera O, Tresserras R, Brugulat P, Mompart A, Medina A, Ferrer M, Alonso J. [Reference guidelines for the 12-Item Short-Form Health Survey version 2 based on the Catalan general population]. Med Clin (Barc). 2012 Dec 8;139(14):613-25. doi: 10.1016/j.medcli.2011.10.024. Epub 2012 Jan 11. Spanish. PMID 22244683
- [Background] Lista-Paz A, Langer D, Barral-Fernandez M, Quintela-Del-Rio A, Gimeno-Santos E, Arbillaga-Etxarri A, Torres-Castro R, Vilaro Casamitjana J, Varas de la Fuente AB, Serrano Veguillas C, Bravo Cortes P, Martin Cortijo C, Garcia Delgado E, Herrero-Cortina B, Valera JL, Fregonezi GAF, Gonzalez Montanez C, Martin-Valero R, Francin-Gallego M, Sanesteban Hermida Y, Gimenez Moolhuyzen E, Alvarez Rivas J, Rios-Cortes AT, Souto-Camba S, Gonzalez-Doniz L. Maximal Respiratory Pressure Reference Equations in Healthy Adults and Cut-off Points for Defining Respiratory Muscle Weakness. Arch Bronconeumol. 2023 Dec;59(12):813-820. doi: 10.1016/j.arbres.2023.08.016. Epub 2023 Sep 29. English, Spanish. PMID 37839949
- [Background] Laveneziana P, Albuquerque A, Aliverti A, Babb T, Barreiro E, Dres M, Dube BP, Fauroux B, Gea J, Guenette JA, Hudson AL, Kabitz HJ, Laghi F, Langer D, Luo YM, Neder JA, O'Donnell D, Polkey MI, Rabinovich RA, Rossi A, Series F, Similowski T, Spengler CM, Vogiatzis I, Verges S. ERS statement on respiratory muscle testing at rest and during exercise. Eur Respir J. 2019 Jun 13;53(6):1801214. doi: 10.1183/13993003.01214-2018. Print 2019 Jun. PMID 30956204
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Gottdiener JS, Bednarz J, Devereux R, Gardin J, Klein A, Manning WJ, Morehead A, Kitzman D, Oh J, Quinones M, Schiller NB, Stein JH, Weissman NJ; American Society of Echocardiography. American Society of Echocardiography recommendations for use of echocardiography in clinical trials. J Am Soc Echocardiogr. 2004 Oct;17(10):1086-119. doi: 10.1016/j.echo.2004.07.013. No abstract available. PMID 15452478
- [Background] Guirao i Goris JA. Elaboración y validación de la versión en español europeo de la escala de valoración rápida de actividad física (RAPA). 2012
- [Background] Topolski TD, LoGerfo J, Patrick DL, Williams B, Walwick J, Patrick MB. The Rapid Assessment of Physical Activity (RAPA) among older adults. Prev Chronic Dis. 2006 Oct;3(4):A118. Epub 2006 Sep 15. PMID 16978493
- [Background] Ambrosetti M, Abreu A, Corra U, Davos CH, Hansen D, Frederix I, Iliou MC, Pedretti RFE, Schmid JP, Vigorito C, Voller H, Wilhelm M, Piepoli MF, Bjarnason-Wehrens B, Berger T, Cohen-Solal A, Cornelissen V, Dendale P, Doehner W, Gaita D, Gevaert AB, Kemps H, Kraenkel N, Laukkanen J, Mendes M, Niebauer J, Simonenko M, Zwisler AO. Secondary prevention through comprehensive cardiovascular rehabilitation: From knowledge to implementation. 2020 update. A position paper from the Secondary Prevention and Rehabilitation Section of the European Association of Preventive Cardiology. Eur J Prev Cardiol. 2021 May 14;28(5):460-495. doi: 10.1177/2047487320913379. PMID 33611446
- [Background] Taylor RS, Brown A, Ebrahim S, Jolliffe J, Noorani H, Rees K, Skidmore B, Stone JA, Thompson DR, Oldridge N. Exercise-based rehabilitation for patients with coronary heart disease: systematic review and meta-analysis of randomized controlled trials. Am J Med. 2004 May 15;116(10):682-92. doi: 10.1016/j.amjmed.2004.01.009. PMID 15121495
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Azambuja ACM, de Oliveira LZ, Sbruzzi G. Inspiratory Muscle Training in Patients With Heart Failure: What Is New? Systematic Review and Meta-Analysis. Phys Ther. 2020 Dec 7;100(12):2099-2109. doi: 10.1093/ptj/pzaa171. PMID 32936904
- [Background] Hossein Pour AH, Gholami M, Saki M, Birjandi M. The effect of inspiratory muscle training on fatigue and dyspnea in patients with heart failure: A randomized, controlled trial. Jpn J Nurs Sci. 2020 Apr;17(2):e12290. doi: 10.1111/jjns.12290. Epub 2019 Aug 19. PMID 31429207
- [Background] Viéitez Flórez JM, Rivas SG, Zamorano Gómez JL. Cardiopatía isquémica: concepto, clasificación, epidemiología, medidas preventivas y tratamiento no farmacológico
- [Background] Fabero-Garrido R, Del Corral T, Plaza-Manzano G, Sanz-Ayan P, Izquierdo-Garcia J, Lopez-de-Uralde-Villanueva I. Effects of Respiratory Muscle Training on Exercise Capacity, Quality of Life, and Respiratory and Pulmonary Function in People With Ischemic Heart Disease: Systematic Review and Meta-Analysis. Phys Ther. 2024 Mar 1;104(3):pzad164. doi: 10.1093/ptj/pzad164. PMID 38015997
- See also: Information about Myocardial Ischemia in the Spanish Heart Foundation website — https://fundaciondelcorazon.com/informacion-para-pacientes/enfermedades-cardiovasculares/cardiopatia-isquemica.html
- See also: Global epidemiology of Ischemia Heart Desease — https://www.cureus.com/articles/36728-global-epidemiology-of-ischemic-heart-disease-results-from-the-global-burden-of-disease-study
- See also: Guidelines of the Spanish Society of Cardiology for Clinical Practice in Exercise Testing — https://www.revespcardiol.org/es-guias-practica-clinica-sociedad-espanola-articulo-X0300893200108041